CLINICAL TRIAL: NCT03843255
Title: Defining the Genetics, Biomarkers and Outcomes for Dilated Cardiomyopathy: a Prospective Multi-centre Observational Study
Brief Title: Defining the Genetics, Biomarkers and Outcomes for Dilated Cardiomyopathy
Acronym: Go-DCM
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: British Heart Foundation (Other); Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18IC4391
Record Dates: First submitted 2019-01-31; First posted 2019-02-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Dilated Cardiomyopathy; Cardiovascular Diseases
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiovascular Diseases | interventions — Whole Genome Sequencing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — 1. Blood- plasma and serum
  2. Saliva
  3. Collection of additional tissue samples (myocardial, skeletal, skin) from planned clinical procedures (where applicable)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Part 1: Dilated Cardiomyopathy patients: Approximately 1200 patients recruited prospectively from participating sites with a diagnosis of Dilated Cardiomyopathy (DCM). Will also include approximately 800 retrospective patients diagnosed with DCM currently biobanked by the lead site.
  Interventions: Other: Part 1: DCM Cohort
- Part 2: Heritable Cardiovascular Disease: Patients may be recruited with other diagnosed heritable cardiovascular disorders. Family members of patients may be invited to take part in the study. Children may also be approached to take part in the study.
  Interventions: Other: Part 2: Heritable CV Diseases and Family Members

INTERVENTIONS:
Other: Part 1: DCM Cohort — Patients with a confirmed diagnosis of DCM will have samples that undergo whole genome sequencing and biomarker analysis
  Other Names: Whole genome sequencing and biomarker analysis
  Groups: Part 1: Dilated Cardiomyopathy patients
Other: Part 2: Heritable CV Diseases and Family Members — Biomarker analysis will be undertaken on samples
  Other Names: Biomarker analysis
  Groups: Part 2: Heritable Cardiovascular Disease

SUMMARY:
Finding new ways to diagnose and treat Dilated Cardiomyopathy (DCM) could improve the health and well-being of patients with this condition. The main aim of this research study is to help develop better ways of diagnosing and treating patients with DCM. The information that is collected may help develop tailored treatments for patients with this disease in the future. This research study will recruit patients with DCM from a number of centres across England and follow their health over a period of years. Patients will give some blood samples for a type of genetic test called whole genome sequencing (WGS) to look for genetic changes. Patients will also have a magnetic resonance imaging (MRI) scan of their heart to look for any changes in the heart such as scarring, and check their heart function. The aim of this study is to discover if using WGS and MRI can improve the diagnosis of DCM. Another aim of the study is to look at how genetic changes and scarring in the heart may affect the progress of the disease.

Studying patients with DCM may also help the investigators learn more about diagnosing and treating other diseases of the heart. The second aim of this study is to see whether using WGS and MRI scanning can also be useful in other types of heart diseases which might be affected by genetic changes or scarring in the heart.

DETAILED DESCRIPTION:
This study will recruit patients from a number of hospitals in England and study them over a number of years. The study will be divided in 2 parts. Part 1 will recruit patients with a diagnosis of DCM, Part 2 will recruit patients diagnosed with other heritable cardiovascular disorders. Family members of patients may be invited to take part in the study. Children may also be approached to take part in the study.

Patients will attend for a baseline visit for a cardiovascular magnetic resonance (CMR) scan, completion of quality of life questionnaires, collection of blood samples for whole genome sequencing and biomarker analysis, and collection of clinical data. Collection of health information via national registries including Office of National Statistics (ONS) and Hospital Episodes Statistics (HES) will be continued over the patients's lifetime. This will not require any direct contact with the participant.

Recruitment will take place over a 3 year period, with annual completion of questionnaires at patients scheduled hospital visits. If the patient is not scheduled to attend the hospital for regular follow up, then patients may complete the questionnaires via an online system or over the telephone. Patients will be asked to complete questionnaires annually for 5 years. Sub-sets of patients may be invited for additional tests including exercise testing, and stress perfusion scans. These tests will not form part of the core tests for the study, and patients may choose not to have them. Separate informed consent will be obtained from participants for any additional tests.

If patients are having clinical diagnostic tests that involve the removal of tissue, they may be asked to donate any surplus tissue sample, or be asked to provide their consent to collect an additional tissue sample. Separate informed consent will be obtained from participants for donation of additional tissue samples.

Where patients are scheduled to have a CMR scan as part of their routine clinical care, an additional CMR scan for research purposes may not be required.

Children will not be asked to complete any annual questionnaires, health information will be collected via ONS and HES.

Family members of patients who take part in the study will only be asked to donate a blood or saliva sample, and provide consent to collection of their health information via ONS and HES records. They will not have any clinical tests such as CMR.

ELIGIBILITY:
PART 1

Inclusion Criteria:

* Male or female participants of any age
* Capacity to provide informed consent
* Patients with a confirmed diagnosis of DCM
* Affected family members of patients meeting diagnostic criteria for DCM

Exclusion Criteria:

* DCM attributed to chemotoxicity (from chemotherapeutic agents, drugs of abuse)
* DCM attributed to systemic inflammatory myopathies (eg sarcoid, systemic lupus erythematosus)
* Patients who lack capacity to consent for themselves
* Patients with a confirmed history of coronary artery disease, assessed using standard UK clinical practice guidelines, defined as one or more of the following:-

  * >50% narrowing, any major epicardial coronary artery on invasive or computed tomography coronary angiography
  * CMR suggestive of previous myocardial infarction of ≥2 segments of ≥50% infarction of the LV wall
  * Previous percutaneous coronary intervention or coronary bypass surgery
* History of primary valvular heart disease or congenital heart disease
* Severe, untreated or untreatable hypertension (systolic blood pressures routinely >180 mm Hg and/or diastolic blood pressures >120 mm Hg)

PART 2

Inclusion Criteria:

* Males or females of any age
* Capacity to provide informed consent
* Patients with hypokinetic non-dilated cardiomyopathy, or
* Family members of DCM patients with possible or probable DCM or
* Patients with a confirmed diagnosis of heritable cardiovascular disease or
* Family members of patients with heritable cardiovascular disease, both affected and unaffected

Exclusion Criteria:

* Patients who lack capacity to consent for themselves
* Patients with a confirmed history of coronary artery disease, assessed using standard UK clinical practice guidelines, defined as one or more of the following:-

  * >50% narrowing, any major epicardial coronary artery on invasive or computed tomography coronary angiography
  * CMR suggestive of previous myocardial infarction of ≥2 segments of ≥50% infarction of the LV wall
  * Previous percutaneous coronary intervention or coronary bypass surgery
* History of primary valvular heart disease or congenital heart disease
* Severe, untreated or untreatable hypertension (systolic blood pressures routinely >180 mm Hg and/or diastolic blood pressures >120 mm Hg)

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients of any age with diagnosed DCM (part 1), and
  * Their family members with other heritable cardiovasacular disease (affected and unaffected), or other eligible patients with hypokinetic non-dilated cardiomyopathy (part 2)
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2027-07-22 (Estimated); Study Completion 2027-07-22 (Estimated)

PRIMARY OUTCOMES:
The incidence of major adverse cardiovascular events over 5 years | 5 years
  The incidence of major adverse cardiovascular events over 5 years,defined as:-
  1. Cardiovascular death
  2. Major arrhythmic events (ventricular fibrillation, unstable sustained ventricular tachycardia, appropriate implantable cardioverter-defibrillator delivered shock, and aborted sudden cardiac death)
  3. Major heart failure events (heart transplantation, left ventricular assist device implantation, unplanned heart failure hospitalisation) We will recruit a group of patients that could be asked to take part in future research projects to evaluate personalised treatments for DCM and other cardiovascular diseases.
Incidence of novel gene variants as assessed using whole genome sequencing | 5 years
  Identifying the gene variants contributing to DCM and specifically the incidence of these variants in the target population.

CONTACTS AND LOCATIONS:
Overall Officials: James Ware, Principal Investigator — Imperial College London
Locations (6):
- United Kingdom (6):
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Glenfield Hospital, Leicester
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - Royal Brompton & Harefield NHS Foundation Trust, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Data dictionaries will be shared with collaborating sites
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: During planning (January 2018) and throughout the study recruitment and follow-up period (Dec 2022)
Access Criteria: Provided through secure data transfer mechanisms approved by Imperial College London and secure email